CLINICAL TRIAL: NCT05123820
Title: A Single-center, Open-label, Two-period, Fixed-sequence Study to Investigate the Effect of a Single Oral Dose of ACT-1014-6470 on the Pharmacokinetics of Omeprazole, Midazolam, and Their Metabolites in Healthy Male Subjects
Brief Title: Pharmacokinetics of Omeprazole and Midazolam When Co-administered With ACT-1014-6470
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ID-087-105; 2021-003615-26 (EudraCT Number)
Record Dates: First submitted 2021-11-05; First posted 2021-11-17 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Drug Drug Interaction; Healthy
Keywords: ACT-1014-6470; Omeprazole; Midazolam
MeSH Terms: interventions — Midazolam; Omeprazole; ACT-1014-6470

STUDY DESIGN:
Intervention Model Description: Two-period, fixed-sequence study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACT-1014-6470, Midazolam and Omeprazole (Experimental): Treatment Period A (Day 1 to Day 2) The plan is that all participants will receive treatment A and then treatment B.
  * A single oral dose of midazolam 2 mg and a single oral dose of omeprazole 20 mg on Day 1.
  Treatment Period B (Day 8 to Day 11)
  * A single oral dose of 100 mg ACT-1014-6470, a single oral dose of 20 mg omeprazole, and a single oral dose of 2 mg midazolam on Day 8.
  Interventions: Drug: Treatment period A; Drug: Treatment period B

INTERVENTIONS:
Drug: Treatment period A — Midazolam solution for oral administration. Omeprazole hard capsule for oral administration.
  Other Names: Midazolam and Omeprazole
Drug: Treatment period B — ACT-1014-6470 soft capsule for oral administration. Midazolam solution for oral administration. Omeprazole hard capsule for oral administration.
  Other Names: ACT-1014-6470, Midazolam and Omeprazole

SUMMARY:
A study on whether ACT-1014-6470 has an effect on how the body takes up, distributes and gets rid of omeprazole and midazolam in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in a language understandable to the participant prior to any study-mandated procedure.
* Healthy male participant aged between 18 and 45 years (inclusive) at Screening.
* Body mass index of 18.5 to 28.0 kg/m2 (inclusive) at Screening.
* Systolic blood pressure 100-140 mmHg, diastolic blood pressure 50-90 mmHg, and pulse rate 45-90 beats per minute (inclusive), measured on either arm, after 5 min in the supine position at Screening and on Day -1.

Exclusion Criteria:

* Previous exposure to ACT-1014-6470.
* Known hypersensitivity to ACT-1014-6470, omeprazole, substituted benzimidazoles, midazolam, or treatments of the same pharmacological classes, or any of their excipients.
* History or clinical evidence of any disease and/or existence of any surgical or medical condition, which in the opinion of the investigator, are likely to interfere with the absorption, distribution, metabolism, or excretion of the study treatment (appendectomy and herniotomy allowed if performed more than 12 weeks prior to administration of [first] study treatment, cholecystectomy not allowed).
* Previous treatment with any prescribed medications (including vaccines [Vaccination regimen against COVID-19 completed less than 2 weeks prior to first study treatment administration or any vaccination against COVID-19 planned before end-of-study]) or over-the-counter (OTC) medications (including herbal medicines such as St John's Wort, homeopathic preparations, vitamins, and minerals) within 3 weeks prior to first study treatment administration.
* Legal incapacity or limited legal capacity at Screening.
* Participant with rare inherited issues of fructose intolerance, glucose-galactose malabsorption, or sucrase-isomaltase insufficiency.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-11-13 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of ACT-1014-6470, midazolam and omeprazole. | Total duration: up to 11 days
  The plasma pharmacokinetic parameters of ACT-1014-6470, midazolam and omeprazole will be derived by non-compartmental analysis of the plasma concentration-time profiles.
Time to reach Cmax (tmax) of ACT-1014-6470, midazolam and omeprazole. | Total duration: up to 11 days
  The plasma pharmacokinetic parameters of ACT-1014-6470, midazolam and omeprazole will be derived by non-compartmental analysis of the plasma concentration-time profiles.
The area under the plasma concentration-time curve (AUC) from zero to time t of the last measured concentration above the limit of quantification (AUC0-t) of ACT-1014-6470, midazolam and omeprazole. | Total duration: up to 11 days
  The plasma pharmacokinetic parameters of ACT-1014-6470, midazolam and omeprazole will be derived by non-compartmental analysis of the plasma concentration-time profiles.
Area under the plasma concentration-time curve [AUC(0-12)] of omeprazole. | Total duration: up to 9 days
  The plasma pharmacokinetic parameters of omeprazole will be derived by non-compartmental analysis of the plasma concentration-time profile.
Area under the plasma concentration-time curve [AUC(0-24)] of midazolam and omeprazole. | Total duration: up to 11 days
  The plasma pharmacokinetic parameters of midazolam and omeprazole will be derived by non-compartmental analysis of the plasma concentration-time profiles.
Area under the plasma concentration-time curve [AUC(0-inf)] of ACT-1014-6470, midazolam and omeprazole. | Total duration: up to 11 days
  The plasma pharmacokinetic parameters of ACT-1014-6470, midazolam and omeprazole will be derived by non-compartmental analysis of the plasma concentration-time profiles.
Apparent total body clearance (CL/F) of ACT-1014-6470, midazolam and omeprazole. | Total duration: up to 11 days
  The plasma pharmacokinetic parameters of ACT-1014-6470, midazolam and omeprazole will be derived by non-compartmental analysis of the plasma concentration-time profiles.
The terminal half-life (t½) of ACT-1014-6470, midazolam and omeprazole. | Total duration: up to 11 days
  The plasma pharmacokinetic parameters of ACT-1014-6470, midazolam and omeprazole will be derived by non-compartmental analysis of the plasma concentration-time profiles.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of 1-hydroxymidazolam and 5-hydroxyomeprazole. | Total duration: up to 11 days
  The plasma pharmacokinetic parameters of 1-hydroxymidazolam and 5-hydroxyomeprazole will be derived by non-compartmental analysis of the plasma concentration-time profiles.
Time to reach Cmax (tmax) of 1-hydroxymidazolam and 5-hydroxyomeprazole. | Total duration: up to 11 days
  The plasma pharmacokinetic parameters of 1-hydroxymidazolam and 5-hydroxyomeprazole will be derived by non-compartmental analysis of the plasma concentration-time profiles.
The area under the plasma concentration-time curve (AUC) from zero to time t of the last measured concentration above the limit of quantification (AUC0-t) of 1-hydroxymidazolam and 5-hydroxyomeprazole. | Total duration: up to 11 days
  The plasma pharmacokinetic parameters of 1-hydroxymidazolam and 5-hydroxyomeprazole will be derived by non-compartmental analysis of the plasma concentration-time profiles.
Area under the plasma concentration-time curve [AUC(0-12)] of 5-hydroxyomeprazole. | Total duration: up to 11 days
  The plasma pharmacokinetic parameters of 5-hydroxyomeprazole will be derived by non-compartmental analysis of the plasma concentration-time profiles.
Area under the plasma concentration-time curve [AUC(0-24)] of 1-hydroxymidazolam and 5-hydroxyomeprazole. | Total duration: up to 11 days
  The plasma pharmacokinetic parameters of 1-hydroxymidazolam and 5-hydroxyomeprazole will be derived by non-compartmental analysis of the plasma concentration-time profiles.
Area under the plasma concentration-time curve [AUC(0-inf)] of 1-hydroxymidazolam and 5-hydroxyomeprazole. | Total duration: up to 11 days
  The plasma pharmacokinetic parameters of 1-hydroxymidazolam and 5-hydroxyomeprazole will be derived by non-compartmental analysis of the plasma concentration-time profiles.
The terminal half-life (t½) of 1-hydroxymidazolam and 5-hydroxyomeprazole. | Total duration: up to 11 days
  The plasma pharmacokinetic parameters of 1-hydroxymidazolam and 5-hydroxyomeprazole will be derived by non-compartmental analysis of the plasma concentration-time profiles.
The metabolic ratio (MR) of 1-hydroxymidazolam to midazolam . | Total duration: up to 11 days
The metabolic ratio (MR) of 5-hydroxyomeprazole to omeprazole. | Total duration: up to 11 days
Number of participants with treatment-emergent adverse events as a measure of safety and tolerability. | Total duration: up to 11 days
  An adverse event is an unfavorable and unintended sign (including an abnormal laboratory finding, an abnormal electrocardiogram). A treatment-emergent adverse event is any adverse event temporally associated with the use of a study treatment, whether or not considered related to the study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- CEPHA s.r.o., Pilsen, Czechia

IPD SHARING:
Plan to Share IPD: No